CLINICAL TRIAL: NCT07344662
Title: The Effect of Hemsball Efficacy on Balance, Kinesiophobic Attitude and Frailty in the Elderly: A Randomized Controlled Trial
Brief Title: The Effect of Hemsball in the Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Şükran İRİBALCI, Assoc.Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SelcukU-SBF-Şİ-02
Record Dates: First submitted 2025-12-30; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Balance; Kinesiophobia; Frailty; Older People; Male; Activities; Hemsball
MeSH Terms: conditions — Kinesiophobia; Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Hemsball group
  Interventions: Other: Experimental: Hemsball
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Experimental: Hemsball — The intervention program was developed within the theoretical framework of the book "Hemsball for All Ages," and expert opinions were sought from both the author of the book and the president of the Hemsball Federation. The program was conducted in groups, and game times were determined for each group. The program continued with groups of five individuals per hour, totaling 10 people, and lasted approximately five hours over half a day with 44 individuals. The older people participants in the Hemsball activity followed the principle of continuity for eight weeks, three days a week, with 60 minutes of Hemsball activity each day.
  Arms: Intervention

SUMMARY:
This study aimed to determine the effect of hemsball activity on balance, kinesiophobic attitudes, and frailty levels in older male individuals. The research was conducted as a parallel-group pre-test-post-test randomized controlled trial. The reporting of the study utilized the CONSORT 2017 extension evaluating non-pharmacological interventions. The study was conducted with 86 older male individuals using a parallel-group pre-test-post-test randomized controlled trial design. The hemsball activity was structured by the research team and lasted for eight weeks, three days a week, for 60 minutes each day. Data were collected using pre-tests planned before randomization, immediately after obtaining written consent from the individuals, and post-tests in the eighth week of the study. Data were collected using a Personal Information Form, the Berg Balance Scale, the Tampa Kinesiophobia Scale, and the Edmonton Frailty Scale. Data were analyzed using a generalized linear model. This research found that hemsball activity is an effective intervention in improving balance and reducing kinesiophobia and frailty in older male individuals. Through this research, a new type of intervention that improves balance and reduces kinesiophobia and frailty levels in older individuals has been added to the literature.

ELIGIBILITY:
Inclusion Criteria:- Being 65 years of age or older being male Having no problems with verbal communication Having no disability including blindness, hearing loss, or limb impairment Having sound mental and psychological health

Exclusion Criteria:

Failing to attend the event three times in a row Having serious chronic illnesses that restrict participation in the event (such as cardiovascular, musculoskeletal, respiratory system diseases..) Having a lower extremity fracture within the last year Having undergone any surgery within the last month Having been diagnosed with any neuropsychiatric disorder (dementia, Alzheimer's disease, traumatic brain injury, Parkinson's disease, stroke, etc.)

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 86 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | It was completed at the beginning of the study and at the end of 8 weeks.
  This form consists of 13 questions designed by researchers to determine individuals' personal characteristics based on the literature.
Berg Balance Scale | at the start of the study and at the end of 8 weeks
  This scale was developed to determine individuals' levels of balance. The scale consists of 14 items, each scored between 0 (poor) and 4 (best). The total score on the scale ranges from 0 to 56. A higher score indicates better balance.
Tampa Kinesiophobia Scale | at the start of the study and at the end of 8 weeks
  This scale assesses individuals' work-related actions, injury/re-injury, and fear-avoidance behaviors. The scale consists of 17 items, scored from 1 (strongly disagree) to 4 (strongly agree). Four items are reverse-scored (items 4, 8, 12, and 16). The total score ranges from 17 to 68. An increased score indicates increased kinesiophobia.
Edmonton Frailty Scale | at the start of the study and at the end of 8 weeks
  This scale assesses the vulnerability of older individuals across dimensions including "cognitive status, general health status, functional independence, social support, medication use, nutrition, mood, urinary incontinence, and functional performance." The scale consists of nine dimensions and 11 items. The total score obtainable from the scale ranges from 0 to 17.

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No